CLINICAL TRIAL: NCT04958226
Title: An Open-label, Fixed-sequence Study to Assess the Effect of Repeated Doses of Capivasertib on the Pharmacokinetics of Oral Midazolam (a CYP450 3A Probe) in Patients With Advanced Solid Tumours
Brief Title: A Study to Assess the Effect of Capivasertib on Midazolam in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D3614C00003
Record Dates: First submitted 2021-07-01; First posted 2021-07-12 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Solid Tumour
Keywords: CYP3A inhibitor; Pharmacokinetics; Safety
MeSH Terms: interventions — capivasertib; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Midazolam + Capivasertib) (Experimental): Midazolam will be administered on Cycle 1 Day 1 and Cycle 1 Day 8. Capivasertib will be administrated from Cycle 1 Day 2 as an intermittent schedule (4 days on/3 days off) until discontinuation. On Cycle 1 Day 12, Midazolam will be administrated with Capivasertib.
  Interventions: Drug: Capivasertib; Drug: Midazolam

INTERVENTIONS:
Drug: Capivasertib — Capivasertib (tablet) will be given as an intermittent schedule (4 days on/3 days off) from Cycle 1 Day 2 until discontinuation. Capivasertib will be administrated in both Part A and Part B.
Drug: Midazolam — Single doses of midazolam (syrup, 1 mg) will be given on cycle 1 Days 1, 8, and 12.

SUMMARY:
This is an open-label, fixed-sequence study to evaluate the effect of capivasertib on the pharmacokinetics (PK) of midazolam, a sensitive CYP3A substrate. The PK of midazolam will be assessed when administered alone and in combination with repeated doses of capivasertib.

DETAILED DESCRIPTION:
This is 2 part study: Part A and Part B. Part A of the study consists of a screening period and 3 treatment periods (midazolam alone, capivasertib alone, and midazolam + capivasertib). During Part A, the PK profile of midazolam will be determined with and without capivasertib.All participants will receive capivasertib treatment (4 days on/3 days off); however, at the Investigator's discretion, ER positive breast cancer patients may also receive fulvestrant in addition to capivasertib and midazolam. Participants completing Part A without disease progression or unacceptable toxicity, who are considered likely to continue to benefit from further capivasertib treatment (with or without certain standard of care treatment) in the opinion of the Investigator will enter Part B. Part B of the study consists of an extended treatment period with capivasertib, with or without certain standard of care treatment, followed by a 30-day safety follow-up.

Part A of the study may be extended to allow the administration of midazolam on a rescheduled Cycle 1 Day 8(C1D8) and Cycle 1 Day 12(C1D12 ) visit.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with documented evidence of locally advanced inoperable or metastatic solid tumours who may be suitable to receive capivasertib treatment.
2. Eastern Cooperative Oncology Group/World Health Organization performance status 0 to 1 and with minimum life expectancy for 12 weeks.
3. Participant should have at least one lesion that can be assessed by computed tomography/magnetic resonance imaging or plain X-ray at baseline.
4. Body mass index within the range 18 to 32 kg/m^2

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Radiotherapy with a wide field of radiation within 4 weeks of the first dose of capivasertib and/or radiotherapy with a limited field of radiation for palliation within 2 weeks prior to study intervention initiation.
2. Participants with diabetes mellitus type I or participants with diabetes mellitus type II requiring insulin treatment.
3. Undergone a major surgery within 4 weeks of the first dose of capivasertib.
4. Any unresolved toxicities from prior therapies higher than CTCAE grade 2 or any unresolved toxicity that may interfere with PK assessment at the time of study intervention initiation.
5. Participants with spinal cord compression or brain metastases.
6. Participants with severe or uncontrolled systemic diseases, active bleeding diatheses, or active infection.
7. Previous allogeneic bone marrow transplant or solid organ transplant.
8. Known immunodeficiency syndrome.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Midazolam AUCinf | Cycle 1 Day 1, Cycle 1 Day 2, Cycle 1 Day 8, Cycle 1 Day 9, Cycle 1 Day 12 and Cycle 1 Day 13 (Cycle 1 is 29 days)
  Area under the plasma concentration-time curve from zero to infinity
Midazolam Cmax | Cycle 1 Day 1, Cycle 1 Day 2, Cycle 1 Day 8, Cycle 1 Day 9, Cycle 1 Day 12 and Cycle 1 Day 13 (Cycle 1 is 29 days)
  Maximum observed plasma (peak) drug concentration

SECONDARY OUTCOMES:
Midazolam AUClast | Cycle 1 Day 1, Cycle 1 Day 2, Cycle 1 Day 8, Cycle 1 Day 9, Cycle 1 Day 12 and Cycle 1 Day 13 (Cycle 1 is 29 days)
  Area under plasma concentration-time curve from zero to the last quantifiable concentration
Midazolam t½λz | Cycle 1 Day 1, Cycle 1 Day 2, Cycle 1 Day 8, Cycle 1 Day 9, Cycle 1 Day 12 and Cycle 1 Day 13 (Cycle 1 is 29 days)
  Half-life associated with terminal slope (λz) of a semilogarithmic concentration-time curve
Midazolam tmax | Cycle 1 Day 1, Cycle 1 Day 2, Cycle 1 Day 8, Cycle 1 Day 9, Cycle 1 Day 12 and Cycle 1 Day 13 (Cycle 1 is 29 days)
  Time to reach peak or maximum observed concentration
Capivasertib Ctrough | Cycle 1 Day 9 and Cycle 1 Day 13 (Cycle 1 is 29 days)
  Observed lowest drug concentration reached before the next dose is administered
Capivasertib Cmax | Cycle 1 Day 12 and Cycle 1 Day 13 (Cycle 1 is 29 days)
  Maximum observed plasma (peak) drug concentration
Capivasertib AUCτ | Cycle 1 Day 12 and Cycle 1 Day 13 (Cycle 1 is 29 days)
  Area under plasma concentration-time curve in the dose interval
Capivasertib t½λz | Cycle 1 Day 12 and Cycle 1 Day 13 (Cycle 1 is 29 days)
  Half-life associated with terminal slope (λz) of a semilogarithmic concentration-time curve
Capivasertib tmax | Cycle 1 Day 12 and Cycle 1 Day 13 (Cycle 1 is 29 days)
  Time to reach peak or maximum observed concentration
Capivasertib CL/F | Cycle 1 Day 12 and Cycle 1 Day 13 (Cycle 1 is 29 days)
  Apparent total body clearance of drug from plasma after extravascular administration
Capivasertib metabolite AZ14102143 Ctrough | Cycle 1 Day 9 and Cycle 1 Day 13 (Cycle 1 is 29 days)
  Observed lowest drug concentration reached before the next dose is administered
Capivasertib metabolite AZ14102143 Cmax | Cycle 1 Day 12 and Cycle 1 Day 13 (Cycle 1 is 29 days)
  Maximum observed plasma (peak) drug concentration
Capivasertib metabolite AZ14102143 AUCτ | Cycle 1 Day 12 and Cycle 1 Day 13 (Cycle 1 is 29 days)
  Area under plasma concentration-time curve in the dose interval
Capivasertib metabolite AZ14102143 t½λz | Cycle 1 Day 12 and Cycle 1 Day 13 (Cycle 1 is 29 days)
  Half-life associated with terminal slope (λz) of a semilogarithmic concentration-time curve
Capivasertib metabolite AZ14102143 tmax | Cycle 1 Day 12 and Cycle 1 Day 13 (Cycle 1 is 29 days)
  Time to reach peak or maximum observed concentration
Number of participants with adverse events and serious adverse events | From screening to disease progression or discontinuation from the study (up to 15 months)
  Assessment of safety and tolerability of capivasertib (with or without the use of standard of care)and in combination with midazolam.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Research Site, Aurora, Colorado
  - Research Site, Durham, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Miller C, Sommavilla R, O'Bryant CL, Barve M, Dowlati A, Luke JJ, Khatun M, Morris T, Cullberg M. Pharmacokinetic study of capivasertib and the CYP3A4 substrate midazolam in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2024 Aug;94(2):223-235. doi: 10.1007/s00280-024-04667-3. Epub 2024 Apr 20. PMID 38643311